CLINICAL TRIAL: NCT00670488
Title: A Phase I Dose Escalation Study of Oral MK-2206 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Dose Escalation Study With MK-2206 in Patients With Locally Advanced or Metastatic Solid Tumors (MK-2206-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2206-002; 2008_513 (Other: Sponsor registry number); MK-2206-002 (Other: Merck Protocol Number)
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-01

CONDITIONS: Locally Advanced Tumors; Metastatic Solid Tumors; Cancer; Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — MK 2206

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- MK-2206 30 mg QOD (Experimental): Participants receive 30 mg oral MK-2206 every other day (QOD) in repeating 4-week treatment cycles.
  Interventions: Drug: MK-2206
- MK-2206 60 mg QOD (Experimental): Participants receive 60 mg oral MK-2206 QOD in repeating 4-week treatment cycles.
  Interventions: Drug: MK-2206
- MK-2206 75 mg QOD (Experimental): Participants receive 75 mg oral MK-2206 QOD in repeating 4-week treatment cycles.
  Interventions: Drug: MK-2206
- MK-2206 90 mg QOD (Experimental): Participants receive 90 mg oral MK-2206 QOD in repeating 4-week treatment cycles.
  Interventions: Drug: MK-2206
- MK-2206 90 mg QW (Experimental): Participants receive 90 mg oral MK-2206 every week (QW) in repeating 4-week treatment cycles.
  Interventions: Drug: MK-2206
- MK-2206 135 mg QW (Experimental): Participants receive 135 mg oral MK-2206 QW in repeating 4-week treatment cycles.
  Interventions: Drug: MK-2206
- MK-2206 200 mg QW (Experimental): Participants receive 200 mg oral MK-2206 QW in repeating 4-week treatment cycles.
  Interventions: Drug: MK-2206
- MK-2206 300 mg QW (Experimental): Participants receive 300 mg oral MK-2206 QW in repeating 4-week treatment cycles.
  Interventions: Drug: MK-2206
- MK-2206 250 mg QW (Experimental): Participants receive 250 mg oral MK-2206 QW in repeating 4-week treatment cycles.
  Interventions: Drug: MK-2206
- MK-2206 150 mg QW (Experimental): Participants receive 150 mg oral MK-2206 QW in repeating 4-week treatment cycles.
  Interventions: Drug: MK-2206

INTERVENTIONS:
Drug: MK-2206 — MK-2206 administered as an oral formulation in rising dose levels on a QOD schedule (30 mg, 60 mg, 75 mg, and 90 mg) or QW schedule (90 mg, 135 mg, 200 mg, 250 mg, and 300 mg) in repeating 4 week cycles, depending upon allocation.

SUMMARY:
The primary purpose of this study is to investigate the Dose Limiting Toxicities (DLTs), pharmacokinetics (PK), and pharmacodynamics (PD) of MK-2206 administered orally to participants with advanced solid tumors. The preliminary efficacy of MK-2206 will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have confirmed locally advanced or metastatic solid tumors that have failed to respond to standard therapy, have gotten worse or have come back after existing therapy
* Has normal organ function; is no greater than 2 on the ECOG Performance Scale
* Has a negative blood or urine pregnancy test within 72 hours of receiving the first dose of study drug if participant is female
* Is able to swallow capsules and has no surgical or bodily condition that will prevent the patient from swallowing and absorbing oral medications on an ongoing basis

Exclusion Criteria:

* Participant has had chemotherapy, radiotherapy, biological therapy or surgery within 4 weeks of starting the study and has not recovered from adverse events caused by the treatment
* Is currently participating or has participated in a study with an investigational compound or device within 30 days
* Has a primary central nervous system tumor
* Has a history or current evidence of heart disease, slow heart rate or untreated high blood pressure
* Is a known diabetic who is taking insulin or oral antidiabetic therapy
* Is pregnant or breastfeeding or planning to become pregnant during the study
* Is HIV-positive
* Has known history of Hepatitis B or C or active Hepatitis A
* Is receiving treatment with oral corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-04-15 (Actual); Primary Completion 2011-07-11 (Actual); Study Completion 2011-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Yap TA, Yan L, Patnaik A, Fearen I, Olmos D, Papadopoulos K, Baird RD, Delgado L, Taylor A, Lupinacci L, Riisnaes R, Pope LL, Heaton SP, Thomas G, Garrett MD, Sullivan DM, de Bono JS, Tolcher AW. First-in-man clinical trial of the oral pan-AKT inhibitor MK-2206 in patients with advanced solid tumors. J Clin Oncol. 2011 Dec 10;29(35):4688-95. doi: 10.1200/JCO.2011.35.5263. Epub 2011 Oct 24. PMID 22025163
- [Derived] Yap TA, Yan L, Patnaik A, Tunariu N, Biondo A, Fearen I, Papadopoulos KP, Olmos D, Baird R, Delgado L, Tetteh E, Beckman RA, Lupinacci L, Riisnaes R, Decordova S, Heaton SP, Swales K, deSouza NM, Leach MO, Garrett MD, Sullivan DM, de Bono JS, Tolcher AW. Interrogating two schedules of the AKT inhibitor MK-2206 in patients with advanced solid tumors incorporating novel pharmacodynamic and functional imaging biomarkers. Clin Cancer Res. 2014 Nov 15;20(22):5672-85. doi: 10.1158/1078-0432.CCR-14-0868. Epub 2014 Sep 19. PMID 25239610

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 104 participants were enrolled and received treatment in this study.
Period: Overall Study
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
Started | 3 | 58 | 3 | 7 | 3 | 5 | 17 | 3 | 3 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 58 | 3 | 7 | 3 | 5 | 17 | 3 | 3 | 2
Not completed — Adverse Event | 0 | 7 | 0 | 3 | 1 | 1 | 5 | 1 | 0 | 1
Not completed — Physician Decision | 1 | 9 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 41 | 3 | 2 | 2 | 4 | 11 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW | Total
Number analyzed (Participants) | 3 | 58 | 3 | 7 | 3 | 5 | 17 | 3 | 3 | 2 | 104
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (9.5) | 58.2 (11.4) | 62.3 (7.6) | 58.0 (13.1) | 59.0 (8.2) | 53.8 (8.8) | 57.9 (13.3) | 58.7 (8.4) | 57.0 (5.6) | 56.0 (18.4) | 58.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 28 | 0 | 4 | 0 | 4 | 7 | 2 | 1 | 1 | 49
  Male | 1 | 30 | 3 | 3 | 3 | 1 | 10 | 1 | 2 | 1 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was any drug-related AE, regardless of grade, leading to a dose modification of MK-2206. Dose-limiting hematologic and nonhematologic toxicities were defined differently and were based on events occurring during the first cycle of study drug administration. Hematologic DLT defined as any Grade (Gr) 4 or greater hematologic toxicity except neutropenia described as follows: Neutropenia that was Gr 4 lasting for ≥7 days, or Gr 3/Gr 4 with fever >38.5°C and/or infection requiring antibiotic or anti-fungal treatment considered DLT. Gr 4 thrombocytopenia (≤25.0 x 10^9/L) was also considered DLT. Non-hematologic DLTs were defined as any Gr 3, 4, or 5 nonhematologic toxicity, with the specific exceptions of: Gr 3 nausea, vomiting, diarrhea, or dehydration occurring with inadequate supportive care and lasting <48 hours; alopecia; inadequately treated hypersensitivity reactions; and Gr 3 elevated transaminases of ≤1 week in duration. A participant could have more than one DLT.
Time Frame: Day 1 to Day 28 (Cycle 1)
Population: The All Participants as Treated (APaT) population: All participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
Number analyzed (Participants) | 3 | 58 | 3 | 7 | 3 | 5 | 17 | 3 | 3 | 2
Participants
  Hyperglycaemia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash | 0 | 5 | 2 | 3 | 0 | 0 | 3 | 2 | 2 | 1
  Rash macular | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stomatitis | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diarrhoea | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pruritis | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Rash generalized | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Dermatitis acneiform | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Total number of participants with DLTs | 0 | 8 | 3 | 4 | 0 | 0 | 4 | 3 | 2 | 1

2. Primary Outcome: Number of Participants With One or More Adverse Events (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition which was temporally associated with the use of the SPONSOR's product, was also an AE. The number of participants that experienced one or more AEs was reported for each dose level group.
Time Frame: Up to 269 days
Population: APaT population: All participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
Number analyzed (Participants) | 3 | 58 | 3 | 7 | 3 | 5 | 17 | 3 | 3 | 2
Participants | 3 | 58 | 3 | 7 | 3 | 5 | 17 | 3 | 3 | 2

3. Primary Outcome: Area Under the Concentration-time Curve of MK-2206 From Time 0 to 48 Hours (AUC0-48hr) in Participants Receiving Multiple QOD Dosing
Description: Blood samples were collected for PK analyses during the first cycle of therapy. Samples were centrifuged, plasma was withdrawn and plasma concentrations were analyzed by high performance liquid chromatography with tandem mass spectroscopy. AUC 0-48hr was calculated for Day 1 and the last day of treatment in Cycle 1 (Day 27) and reported for all dose levels receiving MK-2206 orally QOD (30, 60, 75, and 90 mg QOD).
Time Frame: Days 1 and 27: predose and 0.5, 1, 2, 3, 4, 6, 10, 24, and 48 hours after MK-2206 dosing
Population: All participants who received MK-2206 orally QOD during Cycle 1 (30, 60, 75, and 90 mg QOD) and had available PK data. Data for the MK-2206 QW dose groups (90, 135, 200, 300, 250, and 150 mg QW) are reported separately.
Measure: Mean (Standard Deviation); unit: nM•hr
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
Number analyzed (Participants) | 3 | 58 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0
nM•hr
  Day 1 | 916 (395) | 1950 (832) | 2110 (782) | 3950 (1920) |  |  |  |  |  |
  Last Day (Day 27): number analyzed (Participants) | 1 | 44 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Last Day (Day 27) | NA (NA) — AUC0-48 hr could not be determined due to insufficient data. | 6160 (2690) | NA (NA) — AUC0-48 hr could not be determined due to insufficient data. | 7970 (5990) |  |  |  |  |  |
Statistical Analysis 1: Comparison: MK-2206 60 mg QOD; The Last Day (Day 27)/Day 1 AUC 0-48 hr Geometric Mean Ratio (GMR) was calculated as follows: Last Day (Day 27) AUC 0-48hr Geometric Mean (GM) ÷ Day 1 AUC 0-48hr GM. AUC 0-48hr GMR for last dose (Day 27) calculated using only data from participants who completed cycle one dosing as scheduled and had sufficient data for calculation; Test type: Other; AUC0-48hr GMR = 3.26
Statistical Analysis 2: Comparison: MK-2206 90 mg QOD; The Last Day (Day 27)/Day 1 AUC 0-48 hr GMR was calculated as follows: Last Day (Day 27) AUC 0-48hr GM ÷ Day 1 AUC 0-48hr GM. AUC 0-48hr GMR for last dose (Day 27) calculated using only data from participants who completed cycle one dosing as scheduled and had sufficient data for calculation; Test type: Other; AUC 0-48hr GMR = 3.18

4. Primary Outcome: Maximum Concentration (Cmax) of MK-2206 in Participants Receiving Multiple QOD Dosing
Description: Blood samples were collected for PK analyses during the first cycle of therapy. Samples were centrifuged, plasma was withdrawn and plasma concentrations were analyzed by high performance liquid chromatography with tandem mass spectroscopy. Cmax was calculated for Day 1 and the last day of treatment in Cycle 1 (Day 27) and reported for all dose levels receiving MK-2206 orally QOD (30, 60, 75, and 90 mg QOD).
Time Frame: Days 1 and 27: predose and 0.5, 1, 2, 3, 4, 6, 10, 24, and 48 hours after MK-2206 dosing
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
Number analyzed (Participants) | 3 | 58 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0
nM
  Day 1 | 33.7 (15.8) | 71.6 (36.3) | 102 (79.9) | 132 (76.5) |  |  |  |  |  |
  Last Day (Day 27): number analyzed (Participants) | 1 | 44 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Last Day (Day 27) | NA (NA) — Cmax could not be determined due to insufficient data. | 176 (77.9) | NA (NA) — Cmax could not be determined due to insufficient data. | 232 (148) |  |  |  |  |  |
Statistical Analysis 1: Comparison: MK-2206 60 mg QOD; The Last Day (Day 27)/Day 1 Cmax GMR was calculated as follows: Last Day (Day 27) Cmax GM ÷ Day 1 Cmax GM. Cmax GMR for last dose (Day 27) calculated using only data from participants who completed cycle one dosing as scheduled and had sufficient data for calculation; Test type: Other; Cmax GMR = 2.59
Statistical Analysis 2: Comparison: MK-2206 90 mg QOD; [analysis description as in outcome 4, analysis 1]; Test type: Other; Cmax GMR = 2.67

5. Primary Outcome: Concentration of MK-2206 After 48 Hours (C48hr) in Participants Receiving Multiple QOD Dosing
Description: Blood samples were collected for PK analyses during the first cycle of therapy. Samples were centrifuged, plasma was withdrawn and plasma concentrations were analyzed by high performance liquid chromatography with tandem mass spectroscopy. C48hr was calculated for Day 1 and the last day of treatment in Cycle 1 (Day 27) and reported for all dose levels receiving MK-2206 orally QOD (30, 60, 75, and 90 mg QOD).
Time Frame: Days 1 and 27: predose and 48 hours after MK-2206 dosing.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
Number analyzed (Participants) | 3 | 58 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0
nM
  Day 1 | 14.1 (5.38) | 30.9 (14.4) | 30.6 (12.0) | 64.1 (28.0) |  |  |  |  |  |
  Last Day (Day 27): number analyzed (Participants) | 1 | 44 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Last Day (Day 27) | 67.9 (NA) — Standard Deviation could not be calculated since the N=1. | 100 (45.6) | 110 (NA) — Standard Deviation could not be calculated since the N=1. | 134 (112) |  |  |  |  |  |
Statistical Analysis 1: Comparison: MK-2206 30 mg QOD; The Last Day (Day 27)/Day 1 C48hr GMR was calculated as follows: Last Day (Day 27) C48hr GM ÷ Day 1 C48hr GM. C48hr GMR for last dose (Day 27) calculated using only data from participants who completed cycle one dosing as scheduled and had sufficient data for calculation; Test type: Other; C48hr GMR = 4.33
Statistical Analysis 2: Comparison: MK-2206 60 mg QOD; [analysis description as in outcome 5, analysis 1]; Test type: Other; C48hr GMR = 3.58

6. Primary Outcome: Time to Maximum Concentration (Tmax) of MK-2206 in Participants Receiving Multiple QOD Dosing
Description: Blood samples were collected for PK analyses during the first cycle of therapy. Samples were centrifuged, plasma was withdrawn and plasma concentrations were analyzed by high performance liquid chromatography with tandem mass spectroscopy. Tmax was calculated for Day 1 and the last day of treatment in Cycle 1 and reported for all dose levels receiving MK-2206 orally QOD (30, 60, 75, and 90 mg QOD).
Time Frame: Days 1 and 27: predose and 0.5, 1, 2, 3, 4, 6, 10, 24, and 48 hours after MK-2206 dosing
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
Number analyzed (Participants) | 3 | 58 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0
hour
  Day 1 | 6.0 [4.0 to 6.0] | 4.0 [2.0 to 24.0] | 6.0 [4.0 to 6.0] | 6.0 [4.0 to 10.0] |  |  |  |  |  |
  Last Day (Day 27): number analyzed (Participants) | 1 | 44 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Last Day (Day 27) | 4.0 [4.0 to 4.0] | 6.0 [3.0 to 24.0] | 10.0 [10.0 to 10.0] | 5.0 [4.0 to 6.0] |  |  |  |  |  |

7. Primary Outcome: Apparent Terminal Half-life (t½) of MK-2206 in Participants Receiving Multiple QOD Dosing
Description: Blood samples were collected for PK analyses on Day 27 of the first cycle of therapy. Samples were centrifuged, plasma was withdrawn and plasma concentrations were analyzed by high performance liquid chromatography with tandem mass spectroscopy. t½ (Harmonic mean ± pseudo SD) was calculated and reported for all dose levels receiving MK-2206 orally QOD (30, 60, 75, and 90 mg QOD).
Time Frame: Day 27: predose and 0.5, 1, 2, 3, 4, 6, 10, 24, and 48 hours after MK-2206 dosing.
Population: All participants who received MK-2206 orally QOD on Day 27 of Cycle 1 (30, 60, 75, and 90 mg QOD) and had available PK data. Data for the MK-2206 QW dose groups (90, 135, 200, 300, 250, and 150 mg QW) are reported separately.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
Number analyzed (Participants) | 1 | 44 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
hour | 62.7 (15.1) | 66.3 (17.0) | 66.2 (4.9) | 65.6 (0) |  |  |  |  |  |

8. Primary Outcome: AUC0-168hr in Participants Receiving Multiple QW Dosing
Description: Blood samples were collected for PK analyses during the first cycle of therapy. Samples were centrifuged, plasma was withdrawn and plasma concentrations were analyzed by high performance liquid chromatography with tandem mass spectroscopy. AUC 0-168 was calculated for Day 1 and the last day of treatment in Cycle 1 and reported for all dose levels receiving MK-2206 orally QW (90, 135, 200, 300, 250, and 150 mg QW).
Time Frame: Days 1 and 22: predose and 2, 4, 6, 10, 24, 48, 96 hours, and 168 hours after MK-2206 dosing
Population: All participants who received MK-2206 orally QW during Cycle 1 (90, 135, 200, 300, 250, and 150 mg QW) and had available PK data. Data for the MK-2206 QOD dose groups (30, 60, 75, and 90 mg QOD) are reported separately.
Measure: Mean (Standard Deviation); unit: nM•hr
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 5 | 17 | 3 | 3 | 2
nM•hr
  Day 1 |  |  |  |  | 6510 (3810) | 12000 (4610) | 16400 (5470) | 27700 (3320) | 14000 (2950) | 20700 (0)
  Last Day (Day 22): number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 4 | 13 | 0 | 1 | 1
  Last Day (Day 22) |  |  |  |  | 10600 (7520) | 20700 (8780) | 23500 (14700) |  | 10700 (NA) — Standard Deviation could not be calculated since the N=1. | 22600 (0)
Statistical Analysis 1: Comparison: MK-2206 135 mg QW; The Last Day/Day 1 AUC 0-168 hr GMR was calculated as follows: Last Day AUC 0-168hr GM ÷ Day 1 AUC 0-48hr GM; Test type: Other; AUC0-168hr GMR = 1.91
Statistical Analysis 2: Comparison: MK-2206 200 mg QW; The Last Day/Day 1 AUC 0-168 hr GMR was calculated as follows: Last Day AUC 0-168hr GM ÷ Day 1 AUC 0-48hr GM; Test type: Other; AUC 0-168hr GMR = 1.54

9. Primary Outcome: Cmax of MK-2206 in Participants Receiving Multiple QW Dosing
Description: Blood samples were collected for PK analyses during the first cycle of therapy. Samples were centrifuged, plasma was withdrawn and plasma concentrations were analyzed by high performance liquid chromatography with tandem mass spectroscopy. Cmax was calculated for Day 1 and the last day of treatment in Cycle 1 and reported for all dose levels receiving MK-2206 orally QW (90, 135, 200, 300, 250, and 150 mg QW).
Time Frame: Days 1 and 22: predose and 2, 4, 6, 10, 24, 48, 96 hours, and 168 hours after MK-2206 dosing
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 5 | 17 | 3 | 3 | 2
nM
  Day 1 |  |  |  |  | 81.7 (42.4) | 199 (98.9) | 264 (75.8) | 466 (123) | 231 (39.1) | 337 (0)
  Last Day (Day 22): number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 4 | 13 | 0 | 1 | 1
  Last Day (Day 22) |  |  |  |  | 153 (98.0) | 352 (210) | 345 (199) |  | 169 (NA) — Standard Deviation could not be calculated since the N=1. | 346 (NA) — Standard Deviation could not be calculated since the N=1.
Statistical Analysis 1: Comparison: MK-2206 135 mg QW; The Last Day/Day 1 Cmax GMR was calculated as follows: Last Day Cmax GM ÷ Day 1 Cmax GM; Test type: Other; Cmax GMR = 1.95
Statistical Analysis 2: Comparison: MK-2206 200 mg QW; The Last Day/Day 1 Cmax GMR was calculated as follows: Last Day Cmax GM ÷ Day 1 Cmax GM; Test type: Other; Cmax GMR = 1.33

10. Primary Outcome: C48hr of MK-2206 in Participants Receiving Multiple QW Dosing
Description: Blood samples were collected for PK analyses during the first cycle of therapy. Samples were centrifuged, plasma was withdrawn and plasma concentrations were analyzed by high performance liquid chromatography with tandem mass spectroscopy. C48hr was calculated for Day 1 and the last day of treatment in Cycle 1 and reported for all dose levels receiving MK-2206 orally QW (90, 135, 200, 300, 250, and 150 mg QW).
Time Frame: Days 1 and 22: predose and 48 hours after MK-2206 dosing
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 5 | 17 | 3 | 3 | 2
nM
  Day 1 |  |  |  |  | 50.9 (38.2) | 90.3 (25.1) | 121 (47.4) | 253 (0) | 103 (19.6) | 155 (0)
  Last Day (Day 22): number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 4 | 13 | 0 | 1 | 1
  Last Day (Day 22) |  |  |  |  | 79.3 (33.7) | 158 (59.2) | 187 (113) |  | 74.8 (0) | 185 (0)
Statistical Analysis 1: Comparison: MK-2206 90 mg QOD; The Last Day/Day 1 C48hr GMR was calculated as follows: Last Day C48hr GM ÷ Day 1 C48hr GM; Test type: Other; C48hr GMR = 1.61
Statistical Analysis 2: Comparison: MK-2206 135 mg QW; The Last Day/Day 1 C48hr GMR was calculated as follows: Last Day C48hr GM ÷ Day 1 C48hr GM; Test type: Other; C48hr GMR = 1.86
Statistical Analysis 3: Comparison: MK-2206 200 mg QW; The Last Day/Day 1 C48hr GMR was calculated as follows: Last Day C48hr GM ÷ Day 1 C48hr GM; Test type: Other; C48hr GMR = 1.49

11. Primary Outcome: Tmax of MK-2206 in Participants Receiving Multiple QW Dosing
Description: Blood samples were collected for PK analyses during the first cycle of therapy. Samples were centrifuged, plasma was withdrawn and plasma concentrations were analyzed by high performance liquid chromatography with tandem mass spectroscopy. Tmax was calculated for Day 1 and the last day of treatment in Cycle 1 and reported for all dose levels receiving MK-2206 orally QW (90, 135, 200, 300, 250, and 150 mg QW).
Time Frame: Days 1 and 22: predose and 2, 4, 6, 10, 24, 48, 96 hours, and 168 hours after MK-2206 dosing
Population: as for outcome 8
Measure: Median (Full Range); unit: hour
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 5 | 17 | 3 | 3 | 2
hour
  Day 1 |  |  |  |  | 6.0 [4.0 to 10.0] | 4.0 [4.0 to 10.0] | 6.0 [4.0 to 10.0] | 4.0 [4.0 to 6.0] | 6.0 [4.0 to 6.0] | 7.0 [4.0 to 10.0]
  Last Day (Day 22): number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 4 | 13 | 0 | 1 | 1
  Last Day (Day 22) |  |  |  |  | 4.0 [4.0 to 4.0] | 5.0 [4.0 to 24.0] | 6.0 [4.0 to 24.0] |  | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]

12. Primary Outcome: t½ of MK-2206 in Participants Receiving Multiple QW Dosing
Description: Blood samples were collected for PK analyses during the first cycle of therapy. Samples were centrifuged, plasma was withdrawn and plasma concentrations were analyzed by high performance liquid chromatography with tandem mass spectroscopy. t½ (Harmonic mean ± pseudo SD) was calculated for the last day of treatment in Cycle 1 and reported for all dose levels receiving MK-2206 orally QW (90, 135, 200, 300, 250, and 150 mg QW).
Time Frame: Day 22: predose and 2, 4, 6, 10, 24, 48, 96 hours, and 168 hours after MK-2206 dosing
Population: All participants who received MK-2206 orally QW on Day 22 of Cycle 1 (90, 135, 200, 300, 250, and 150 mg QW) and had available PK data. Data for the MK-2206 QOD dose groups (30, 60, 75, and 90 mg QOD) are reported separately.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 4 | 13 | 0 | 1 | 1
hour |  |  |  |  | 71.6 (12.2) | 88.9 (26.9) | 75.1 (14.7) |  | 53.7 (0) | 64.4 (0)

13. Secondary Outcome: Phosphorylated Protein Kinase B (pAkt) Level on Cycle 1 Day 15 (C1D15) After Treatment With MK-2206 at the Maximum Tolerated Dose (MTD)
Description: To determine the inhibition of pAkt by MK-2206 in participants treated at the MTD, levels of Akt phosphorylated at the serine 473 residue (pAkt Ser473 Akt) were measured in snap-frozen tumors collected at baseline and Day 15 of Cycle 1 using a MesoScale enzyme-linked immunosorbent assay (ELISA). Per protocol, pAkt levels were determined only for the MK-2206 MTD (60 mg QOD) group.
Time Frame: Baseline, Cycle 1 Day 15
Population: Participants treated at the MTD (60 mg QOD) dose level with measurable disease at baseline per RECIST and paired tumor samples at baseline and C1D15. Per protocol, no other dose level groups were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: pAkt lysate units/mg protein
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
Number analyzed (Participants) | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
pAkt lysate units/mg protein
  Baseline |  | 2.15 [0.43 to 10.49] |  |  |  |  |  |  |  |
  Cycle 1 Day 15 |  | 0.29 [0.13 to 0.64] |  |  |  |  |  |  |  |
Statistical Analysis 1: Comparison: MK-2206 60 mg QOD; pAkt Geometric Mean Ratio (GMR) = Day 15 Geometric Mean (GM) ÷ Baseline GM; Test type: Other; GMR = 0.133, 95% CI 2-sided [0.051 to 0.347]

14. Secondary Outcome: Number of Participants With Confirmed Response as Per Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Overall tumor response was assessed during the study by diagnostic anatomic imaging using RECIST. The number of participants with a confirmed Complete Response (CR: Disappearance of all target lesions) as per RECIST was reported for each dose level group.
Time Frame: From Cycle 1 Day 1 through the End of Study Visit (up to 6 months)
Population: All participants with measurable disease at baseline per RECIST.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
Number analyzed (Participants) | 3 | 58 | 3 | 7 | 3 | 5 | 17 | 3 | 3 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 269 days
Description: APaT population: All participants who received at least one dose of study treatment.
Arm/Group | MK-2206 30 mg QOD | MK-2206 60 mg QOD | MK-2206 75 mg QOD | MK-2206 90 mg QOD | MK-2206 90 mg QW | MK-2206 135 mg QW | MK-2206 200 mg QW | MK-2206 300 mg QW | MK-2206 250 mg QW | MK-2206 150 mg QW
All-Cause Mortality (participants affected / at risk) | 0/3 | 5/58 | 0/3 | 0/7 | 0/3 | 2/5 | 3/17 | 0/3 | 0/3 | 1/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 21/58 | 0/3 | 5/7 | 0/3 | 3/5 | 8/17 | 2/3 | 0/3 | 2/2
Other Adverse Events (participants affected / at risk) | 3/3 | 56/58 | 3/3 | 7/7 | 3/3 | 4/5 | 16/17 | 3/3 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2206 30 mg QOD (N=3) | MK-2206 60 mg QOD (N=58) | MK-2206 75 mg QOD (N=3) | MK-2206 90 mg QOD (N=7) | MK-2206 90 mg QW (N=3) | MK-2206 135 mg QW (N=5) | MK-2206 200 mg QW (N=17) | MK-2206 300 mg QW (N=3) | MK-2206 250 mg QW (N=3) | MK-2206 150 mg QW (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
QRS axis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (2)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular compression (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2206 30 mg QOD (N=3) | MK-2206 60 mg QOD (N=58) | MK-2206 75 mg QOD (N=3) | MK-2206 90 mg QOD (N=7) | MK-2206 90 mg QW (N=3) | MK-2206 135 mg QW (N=5) | MK-2206 200 mg QW (N=17) | MK-2206 300 mg QW (N=3) | MK-2206 250 mg QW (N=3) | MK-2206 150 mg QW (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lens disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Maculopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Optic disc disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 10 (15) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 8 (11) | 1 (1) | 4 (6) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 22 (31) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 7 (9) | 1 (1) | 0 (0) | 1 (4)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral mucosal exfoliation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 5 (8) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 16 (28) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (4)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (2) | 26 (34) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 8 (10) | 1 (1) | 2 (2) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 4 (6) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 5 (10) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 16 (22) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 8 (17) | 2 (2) | 2 (2) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (10) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 9 (10) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sensory loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (7) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (11) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 26 (41) | 3 (5) | 4 (4) | 0 (0) | 2 (2) | 5 (13) | 3 (8) | 2 (5) | 2 (3)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.